CLINICAL TRIAL: NCT03643094
Title: Golden Black Seed: Support of Metabolic Health and General Wellness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Collaborators: New Chapter Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 044-031
Record Dates: First submitted 2018-03-13; First posted 2018-08-22 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2018-03

CONDITIONS: Hyperlipidemias; Hyperglycemia
MeSH Terms: conditions — Hyperlipidemias; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Open-labeled 8-week study design with evaluation at baseline, 4, and 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golden Black Seed (Experimental): Golden Black Seed, 1 capsule per day for 8 weeks.
  Interventions: Dietary Supplement: Golden Black Seed

INTERVENTIONS:
Dietary Supplement: Golden Black Seed — 1 capsule per day for 8 weeks.

SUMMARY:
To document effects of consuming Golden Black Seed (brand: New Chapter Inc.) on metabolic health and wellness in human subjects.

Golden Black Seed contains extracts from the turmeric root (Curcuma longa) and black cumin seeds (Nigella sativa). Both botanicals have been used traditionally in Asian cooking, and also in herbal medicine for reducing inflammation.

DETAILED DESCRIPTION:
For this clinical study, human participants will be tested over a period of 8 weeks. Below is a simplified diagram illustrating the involvement of each human subject, where all study participants will be tested on three different clinic days.

ELIGIBILITY:
Inclusion Criteria:

1. Adult people of either gender;
2. Age 40-75 years (inclusive);
3. BMI 25-34.9 (inclusive);

Exclusion Criteria:

1. Cancer during past 12 months;
2. Chemotherapy during past 12 months;
3. Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery is allowed, including previous removal of appendix and gall bladder);
4. Currently consuming large doses of anti-inflammatory nutritional supplements, and unwilling to stop taking these supplements for 2 weeks prior to and during the study;
5. Use of oral, inhaled or injected steroid medication within the last 6 months (for example: prednisone, dexamethasone). Nasal sprays for allergies are allowed;
6. Active uncontrolled auto-immune disease (for example: rheumatoid arthritis, lupus, inflammatory bowel disease, Celiac disease);
7. Currently experiencing intense stressful events or life changes;
8. Currently in intensive athletic training (such as marathon runners);
9. Women of childbearing potential, who are pregnant, nursing, or trying to become pregnant;
10. Known food allergies or sensitivities related to the test products or placebo;
11. History of drug abuse during past two years;
12. Participation in another clinical trial involving a consumable test product.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline cholesterol at 8 weeks. | 8 weeks
  Cholesterol levels will be measured at baseline and after 8 weeks.

SECONDARY OUTCOMES:
Change from baseline Superoxide Dismutase at 8 weeks. | 8 weeks
  Superoxide dismutase will be measured at baseline and after 8 weeks.
Change from baseline lipid peroxidation at 8 weeks. | 8 weeks
  Lipid peroxidation will be measured at baseline and after 8 weeks.
Change from baseline 8-OHdG marker for oxidative DNA damage at 8 weeks. | 8 weeks
  8-OHdG will be measured at baseline and after 8 weeks.
Change from baseline fasting glucose at 8 weeks. | 8 weeks
  Fasting glucose will be measured at baseline and after 8 weeks.
Change from baseline leptin at 8 weeks. | 8 weeks
  Leptin will be measured at baseline and after 8 weeks.

OTHER OUTCOMES:
Change from baseline Wellness at 8 weeks. | 8 weeks
  Wellness Questionnaire will be administered at baseline and 8 weeks (scales 0-10)
Change from baseline body composition at 8 weeks. | 8 weeks
  Dexa scan for fat mass (kg) will be performed at baseline and 8 weeks.
Change from baseline blood pressure at 8 weeks. | 8 weeks
  Blood pressure will be measured at baseline and after 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Gitte Jensen, Klamath Falls, Oregon, United States